CLINICAL TRIAL: NCT06696989
Title: Comparative Effects of Frenkel's and Core Stability Exercises on Coordination and Balance in Children With Cerebral Palsy
Brief Title: Comparative Effects of Frenkel's and Core Stability Exercises in Children With Cerebral Palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0240
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Core Stability; Balance; Frenkel exercises
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( Frenkel's exercises) (Experimental): In this group, participants will receive Frenkel's exercises for the lower limb in lying, sitting, and standing positions. And for the upper limb.
  Interventions: Other: Frenkel's exercises
- Group B (Core Stability Exercises) (Experimental): Participants will receive core stability exercises, i.e., abdominal draw-in, roll-up, superman, and bridging.
  Interventions: Other: Core stability exercises

INTERVENTIONS:
Other: Frenkel's exercises — In this group, participants will receive Frenkel's exercises, and the total treatment session will be 60 minutes of routine physical therapy, i.e., breathing, stretching, ROM's, and joint mobility, with rest intervals in between for 20 minutes. To begin the intervention, the investigator will perform Frenkel's exercises for 40 minutes in total, with rest intervals between each exercise, initially performing 5 repetitions and then gradually progressing to 10 and then 15 repetitions, respectively, after 2 weeks.
  Arms: Group A ( Frenkel's exercises)
Other: Core stability exercises — This group participants will receive core stability exercises, and the total treatment session will also be 60 minutes. The routine physical therapy includes breathing, stretching, joint rotations, ROM's, and frequent periods of rest in between the treatment sessions. To begin the intervention the investigator will perform core stability exercises for 40 minutes in total with rest intervals between each exercise and initially performing 5 repetitions and then gradually progressing to 10 and then 15 repetitions, respectively after 2 weeks.
  Arms: Group B (Core Stability Exercises)

SUMMARY:
The aim of this study is to determine and compare the effects of Frenkel's and core stability exercises on the motor function, postural stability and core muscle strength in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a brain injury that manifests as a mobility and posture impairment in infancy or early childhood. Frenkel exercises are series of movements with increasing difficulty that can be performed by ataxic patients in order to regain coordinated, smooth and rhythmic movement. The Core stability Exercises are for the spine, pelvis, and kinetic chain to all balance properly under stress, core stability is necessary. The aim of this study is to determine and compare the effects of Frenkel's and core stability exercises on the motor function, postural stability and core muscle strength in children with cerebral palsy. This will be a Randomized Clinical Trial in which 50 participants with cerebral palsy will be included as per sample size calculation through non probability convenience sampling technique. The study will be single blinded. Participants that achieve the required standards of inclusion and exclusion criteria will be randomly allocated using online randomization tool into two Groups. Group A will receive Frenkel's exercises and Group B will receive core stability exercises, both groups will receive the treatment for 40 minutes with the routine physical therapy for 20 minutes and short-term rest intervals in between for 3 alternative days per week for 12 weeks. Participants initial screening will be done through Gross Motor Function Classification System (GMFCS). The balance will be assessed through the Pediatric Balance Test (PBS), coordination will be assessed through Finger and Nose Test, Heel Shin Test, Catching and Throwing Tasks.

ELIGIBILITY:
Inclusion Criteria:

* The participants fulfilling the given criteria will be included.
* Age: 6 To 12 Years
* Gender: Both male and female
* Children with ataxic cerebral palsy
* Children having level II and III on Gross Motor Functional Classification System (GMFCS)
* Children able to understand the test instruction, able to sit and stand.
* Children with and without using Botulinum Toxin Injections
* The Pediatric Balance Scale (PBS) of 54.6

Exclusion Criteria:

* Severe Cognitive Dysfunction
* Visual problems
* Vestibular Dysfunction
* Uncontrolled epilepsy
* Severe Orthopedic Condition affecting Lower limbs Mobility

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Finger to nose test | 12th week
  The Finger-to-Nose Test measures smooth, coordinated upper-extremity movement by having the examinee touch the tip of his or her nose with his or her index finger. Evaluation of coordination with the Finger-Nose Test is an essential part of the neurological examination
Heel shin test | 12th week
  The heel-shin test is a part of the neurological examination of coordination: the patient runs the sole of one foot up and down the shin of the opposite leg.
Catching and throwing tasks | 12th week
  Ball catching is a skill included in most tests for assessing the motor impairment of children with a mild motor deficit. To objectively measure ball catching short and long ball catching tests were developed to assess children between seven and nine years of age
PBS (Pediatric Ballance Scale) | 12th week
  A modified version of the Berg Balance Scale, the Pediatric Balance Scale is used to evaluate school-age children's functional balance abilities. The 14 items on the scale have a maximum score of 56 points and are rated from 0 (lowest function) to 4 (highest function).

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd, Principal Investigator — Riphah International University
Locations (1):
- RehabCure, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Hlaing SS, Puntumetakul R, Khine EE, Boucaut R. Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 30;22(1):998. doi: 10.1186/s12891-021-04858-6. PMID 34847915
- [Background] Abd-Elfattah HM, Aly SM. Effect of Core Stability Exercises on Hand Functions in Children With Hemiplegic Cerebral Palsy. Ann Rehabil Med. 2021 Feb;45(1):71-78. doi: 10.5535/arm.20124. Epub 2021 Feb 9. PMID 33557483
- [Background] Ali MS, Awad AS, Elassal MI. The effect of two therapeutic interventions on balance in children with spastic cerebral palsy: A comparative study. J Taibah Univ Med Sci. 2019 Jul 26;14(4):350-356. doi: 10.1016/j.jtumed.2019.05.005. eCollection 2019 Aug. PMID 31488967
- [Background] Manko G, Pieniazek M, Tim S, Jekielek M. The Effect of Frankel's Stabilization Exercises and Stabilometric Platform in the Balance in Elderly Patients: A Randomized Clinical Trial. Medicina (Kaunas). 2019 Sep 11;55(9):583. doi: 10.3390/medicina55090583. PMID 31514453
- [Background] Horber V, Fares A, Platt MJ, Arnaud C, Krageloh-Mann I, Sellier E. Severity of Cerebral Palsy-The Impact of Associated Impairments. Neuropediatrics. 2020 Apr;51(2):120-128. doi: 10.1055/s-0040-1701669. Epub 2020 Mar 2. PMID 32120428
- [Background] Graham D, Paget SP, Wimalasundera N. Current thinking in the health care management of children with cerebral palsy. Med J Aust. 2019 Feb;210(3):129-135. doi: 10.5694/mja2.12106. Epub 2019 Feb 10. PMID 30739332
- [Background] Paul S, Nahar A, Bhagawati M, Kunwar AJ. A Review on Recent Advances of Cerebral Palsy. Oxid Med Cell Longev. 2022 Jul 30;2022:2622310. doi: 10.1155/2022/2622310. eCollection 2022. PMID 35941906
- [Background] Khan SA, Talat S, Malik MI. Risk factors, types, and neuroimaging findings in Children with Cerebral Palsy. Pak J Med Sci. 2022 Sep-Oct;38(7):1738-1742. doi: 10.12669/pjms.38.7.6175. PMID 36246690